CLINICAL TRIAL: NCT03134482
Title: Comparison of Clinical Outcomes Between in Vitro Maturation and Minimal Stimulation in Vitro Fertilization in Patients With Polycystic Ovarian Syndrome; Prospective, Randomized Controlled, Parallel, Open-label, Clinical Trial
Brief Title: Comparison of Clinical Outcomes Between IVM and Minimal Stimulation IVF in Patients With PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, You Shin Kim, Associate professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chau
Record Dates: First submitted 2017-04-11; First posted 2017-05-01 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: No Condition
Keywords: in vitro maturation (IVM); polycystic ovarian syndrome (PCOS); ovarian hyperstimulation syndrome (OHSS); assisted reproductive technology (ART)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In vitro maturation (IVM) (Experimental): hCG primed in vitro maturation (IVM) procedure Gonadotropin is not used in this patient group If the endometrial thickness in 6mm or more and the mean diameter of largest follicle is 11 mm or less on menstrual cycle day 9 to 12 on ultrasonography, oocyte retrieval is planned two days later.
  Recombinant hCG injection (priming) is given 36 hour before oocyte retrieval, followed by intracytoplasmic sperm injection (ICSI) for oocyte fertilization.
  The biochemical pregnancy is confirmed by serum beta hCG 15 days later oocyte retrieval.
  The clinical pregnancy is confirmed when gestational sac is detected by transvaginal ultrasonography 3 weeks later oocyte retrieval.
  Interventions: Procedure: IVM
- Minimal stimulation IVF (Active Comparator): minimal stimulation IVF procedure These patients are stimulated with 150 or less IU of recombinant Follicle-stimulating hormone (FSH) from menstrual cycle day 3 in GnRH antagonist protocol.
  If the mean diameters of two or more follicles are 17mm or more, oocyte retrieval is planned two days later.
  Recombinant hCG is triggered 36 hour before oocyte retrieval, followed by intracytoplasmic sperm injection (ICSI) for oocyte fertilization if needed.
  The biochemical pregnancy is confirmed by serum beta hCG 14 days later oocyte retrieval.
  The clinical pregnancy is confirmed when gestational sac is detected by transvaginal ultrasonography 3 weeks later oocyte retrieval.
  Interventions: Procedure: Minimal stimulation IVF

INTERVENTIONS:
Procedure: IVM — No gonadotropin is used, but hCG priming is utilized 36 hour before oocyte maturation.
  Arms: In vitro maturation (IVM)
Procedure: Minimal stimulation IVF — IVF with minimal use of gonadotropin, i.e. 150 or less IU of recombinant FSH, followed by hCG triggering in GnRH antagonist protocol.
  Arms: Minimal stimulation IVF

SUMMARY:
Polycystic ovarian syndrome (PCOS) is most common endocrinologic disease in women of reproductive age with incidence of 6.6 ~ 8%. About fifty percent of the patients with PCOS manifest subfertility and significant proportion of these woman need assisted reproductive technology (ART). These patients are very sensitive to gonadotropins during conventional in vitro fertilization (IVF) and the risk of ovarian hyperstimulation syndrome (OHSS) is high. In vitro maturation (IVM) is an emerging alternative option to conventional IVF for minimizing the risk of OHSS in patients with PCOS. Until now, several studies has been reported the favorable outcomes of oocyte maturation rate, fertilization rate, clinical pregnancy rate, and live birth rate during IVM procedure. However, these results were from retrospective or observational study and there was no suitable randomized controlled trial (RCT).

Therefore, this prospective RCT is aimed to compare and analyze the clinical outcomes between IVM and minimal stimulation IVF in women with PCOS, assessing if IVM is recommendable clinical practice or not.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is most common endocrinologic disease in women of reproductive age with incidence of 6.6 ~ 8%. About fifty percent of the patients with PCOS manifest subfertility and significant proportion of these women need assisted reproductive technology (ART). These patients are very sensitive to gonadotropins during conventional in vitro fertilization (IVF) and the risk of ovarian hyperstimulation syndrome (OHSS), an iatrogenic complication, is very high.

In vitro maturation (IVM) is has been suggested as an alternative option to conventional IVF for eliminating the risk of OHSS in patients with PCOS. In 1994, Trounson et al succeeded in fertilization of in vitro matured oocytes and transferring embryo during unstimulated IVF procedure in women with PCOS. Since then IVM was developed as one method of ART field.

Previously it had been reported that maturation rate of oocytes retrieved from patients with PCOS were lower than oocytes from women without PCOS. However, in several observational studies, maturation rate of oocytes was up to 80.3%, fertilization was up to 21.9%~50% per cycle, and live birth rated was 15.9% per retrieval and 33% per cycle. And in several retrospective case-control studies of comparing IVM and conventional IVF, the miscarriage rate and ectopic pregnancy rate were similar, whereas the maturation rate of oocyte was up to 84%, fertilization rate was 43~70% and pregnancy rate was 22~56%. Because ovarian stimulation is not utilized, OHSS risk is preventable and cost is effective in IVM procedure.

Generally there are three types of IVM techniques; firstly, gonadotropin priming, in which technique small amount of gonadotropin is used for 3 to 5 days. Secondly, human chorionic gonadotropin (hCG) priming, in which hCG is used before oocyte retrieval. Thirdly, no gonadotropin and hCG priming is used. In gonadotropin-priming IVM technique, it had been reported that the number of retrieved oocytes were increased and pregnancy rate was improved from 0 to 29%, but there was no clear evidence of the efficacy. hCG priming technique, most commonly used technique, is for promoting meiotic resumption before full maturation of oocyte. The maturation rate of oocytes was 69~84%, fertilization rate 45 ~ 80%, pregnancy rate 31 ~ 38.5% and live birth rate was 33% in the studies of investigating hCG priming IVM technique in women with PCOS.

Summarizing these observational and retrospective studies, it is expectable that IVM is promising ART method in patients with PCOS, minimizing the risk of OHSS with improved clinical pregnancy rate. However, there was no suitable randomized controlled trial (RCT) to confirm whether IVM is recommendable primary clinical ART practice to women with PCOS.

Therefore, this prospective RCT is aimed to compare and analyze the clinical outcomes between hCG-primed IVM protocol and minimal stimulation IVF with Gonadotropin-releasing hormone (GnRH) antagonist protocol in women with PCOS in fresh cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS under age of 40 years (PCOS diagnosis is based on Revised 2003 Rotterdam criteria of PCOS)

Exclusion Criteria:

* severe male factor subfertility requiring testicular sperm extraction (TESE) or oligoasthenoteratozoospermia
* couples requiring preimplantation genetic screening or diagnosis
* women had undergone ovarian stimulation 30 days before assisted reproductive technology (ART)
* women with severe endometriosis or dysfunctional uterine bleeding
* women with severe uterine factor subfertility (ex. submucosal myoma, intramural myoma protruding endometrium, severe intrauterine adhesion, etc)
* women with ovarian malignancy
* women with severe tubal factor subfertility (ex. persistent hydrosalpinx even after surgery)
* women had undergone treatment of malignancy 5 years before screening of this trial
* women with history of thromboembolism
* women with age of 40 years or more
* women with stimulation dose over 150 IU of exogenous FSH

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | At 6 weeks of pregnancy
  Clinical pregnancy was determined by observation of a gestational sac with fetal heart beat by transvaginal ultrasound scan.

SECONDARY OUTCOMES:
Incidence rate of Ovarian hyperstimulation syndrome (OHSS) | Until three weeks later after hCG injection
  OHSS rate in each arm. Patients' symptoms (abdominal distension, bloating and pain, nausea, vomiting, palpitation) and ultrasonographic findings (fluid collection in pelvic and abdominal cavity, enlarged ovarian size) are investigated for OHSS detection.

CONTACTS AND LOCATIONS:
Overall Officials: You Shin Kim, MD, PhD, Principal Investigator — Fertility center of CHA Gangnam medical center, CHA university
Locations (2):
- South Korea (2):
  - CHA Fertility Center, Seoul station, Seoul
  - CHA Gangnam medical center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siristatidis CS, Vrachnis N, Creatsa M, Maheshwari A, Bhattacharya S. In vitro maturation in subfertile women with polycystic ovarian syndrome undergoing assisted reproduction. Cochrane Database Syst Rev. 2013 Oct 8;(10):CD006606. doi: 10.1002/14651858.CD006606.pub3. PMID 24101529
- [Background] Cha KY, Chung HM, Lee DR, Kwon H, Chung MK, Park LS, Choi DH, Yoon TK. Obstetric outcome of patients with polycystic ovary syndrome treated by in vitro maturation and in vitro fertilization-embryo transfer. Fertil Steril. 2005 May;83(5):1461-5. doi: 10.1016/j.fertnstert.2004.11.044. PMID 15866585
- [Background] Choi MH, Lee SH, Kim HO, Cha SH, Kim JY, Yang KM, Song IO, Koong MK, Kang IS, Park CW. Comparison of assisted reproductive technology outcomes in infertile women with polycystic ovary syndrome: In vitro maturation, GnRH agonist, and GnRH antagonist cycles. Clin Exp Reprod Med. 2012 Dec;39(4):166-71. doi: 10.5653/cerm.2012.39.4.166. Epub 2012 Dec 31. PMID 23346527
- [Background] Child TJ, Phillips SJ, Abdul-Jalil AK, Gulekli B, Tan SL. A comparison of in vitro maturation and in vitro fertilization for women with polycystic ovaries. Obstet Gynecol. 2002 Oct;100(4):665-70. doi: 10.1016/s0029-7844(02)02193-2. PMID 12383531
- [Background] Chian RC, Buckett WM, Tulandi T, Tan SL. Prospective randomized study of human chorionic gonadotrophin priming before immature oocyte retrieval from unstimulated women with polycystic ovarian syndrome. Hum Reprod. 2000 Jan;15(1):165-70. doi: 10.1093/humrep/15.1.165. PMID 10611207
- [Background] Soderstrom-Anttila V, Makinen S, Tuuri T, Suikkari AM. Favourable pregnancy results with insemination of in vitro matured oocytes from unstimulated patients. Hum Reprod. 2005 Jun;20(6):1534-40. doi: 10.1093/humrep/deh768. Epub 2005 Feb 3. PMID 15695312
- [Background] Reavey J, Vincent K, Child T, Granne IE. Human chorionic gonadotrophin priming for fertility treatment with in vitro maturation. Cochrane Database Syst Rev. 2016 Nov 16;11(11):CD008720. doi: 10.1002/14651858.CD008720.pub2. PMID 27852101
- [Background] Aboulghar MA, Mansour RT. Ovarian hyperstimulation syndrome: classifications and critical analysis of preventive measures. Hum Reprod Update. 2003 May-Jun;9(3):275-89. doi: 10.1093/humupd/dmg018. PMID 12859048
- [Derived] Siristatidis CS, Papapanou M, Maheshwari A, Vaidakis D. In vitro maturation in subfertile women with polycystic ovarian syndrome undergoing assisted reproduction. Cochrane Database Syst Rev. 2025 Feb 6;2(2):CD006606. doi: 10.1002/14651858.CD006606.pub5. PMID 39912435